CLINICAL TRIAL: NCT03912961
Title: Comparative Analysis of Diabetic Retinopathy Images by Retina Specialists Versus EyeStar's Artificial Intelligence Software of Images Captured by Pictor Plus Retinal Camera
Brief Title: The Santa Cruz Diabetic Retinopathy Utilizing Artificial Intelligence Study
Acronym: SC-DRAI
Status: Completed | Type: Observational
Sponsor: Retina Global (Other)
Collaborators: VisionQuest Biomedical LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-BOL-SC-DRAI
Record Dates: First submitted 2019-03-13; First posted 2019-04-11 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Picture of the retina with a handheld retinal camera — Patient with diabetes will have their undilated and dilated images taken, with the images being centered on the macula and on the optic disc.

SUMMARY:
In this clinical trial, we plan to evaluate the usefulness of artificial intelligence (AI) software paired with a handheld retinal camera to compare diabetic retinopathy status in Bolivian patients as read by retina specialists versus the AI software.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects who are at least 18 years old who have full legal capacity to volunteer on the date the informed consent is signed;
2. Subjects who can follow the instructions by the clinical staff at the clinical site, and can attend examinations on the scheduled examination dates;
3. Subjects who have been diagnosed with Type I or Type II diabetes mellitus.

Exclusion Criteria:

1. Subjects unable to tolerate ophthalmic imaging;
2. Subjects who have been scheduled for but have not yet undergone the following surgeries: Cataract Surgery (including any related follow-up procedures) or Vitrectomy.
3. Subject blind in one eye due to any cause
4. Subjects who have a condition or a situation, which in the investigator's opinion, may put the subject at increased risk, confound study data, or interfere significantly with the subject's study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are known diabetics in the hospital, or seeking help from the eye clinics or from associated specialties, e.g. endocrinology, will be included in the study as subjects. The Investigators will also recruit subjects who are evaluated in organized outreach visits in the community.
Sampling Method: Non-Probability Sample
Enrollment: 1034 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-04-14 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Number of subjects where the image readout by retina specialists match the readouts by EyeStar AI system for identifying diabetic eye disease | 3 months
  To quantify image analysis performance of the EyeStar AI system paired with Pictor Plus cameras for the detection of referable Diabetic Retinopathy (DR), defined as severe non-proliferative diabetic retinopathy (NPDR), proliferative diabetic retinopathy (PDR), or diabetic macular edema (DME) against adjudicated reads of retinal images by retina specialists

SECONDARY OUTCOMES:
Number of subjects with gradable images taken by the hand held camera | 3 months
  Pictures taken by the handheld retinal camera will be graded by the retina specialists for the quality of image for readouts
Number of subjects with ocular diseases other than diabetic retinopathy between the readout by the EyeStar AI system and those by the retina specialists | 3 months
  To assess the performance of the system in detection of other ocular diseases such as macular degeneration and glaucoma

CONTACTS AND LOCATIONS:
Overall Officials: Rajat Agrawal, MD MS, Study Director — Retina Global
Locations (3):
- Bolivia (3):
  - Centro Medico Kolping, Santa Cruz de la Sierra
  - Clinica Incor, Santa Cruz de la Sierra
  - Hospital Universitario Japones, Santa Cruz de la Sierra

IPD SHARING:
Plan to Share IPD: No